CLINICAL TRIAL: NCT02782741
Title: A Phase 3 Randomized, Multicenter, Multinational, Double-blinded Study Comparing the Efficacy and Safety of Repeated Biweekly Infusions of Avalglucosidase Alfa (neoGAA, GZ402666) and Alglucosidase Alfa in Treatment naïve Patients With Late-onset Pompe Disease
Brief Title: Study to Compare the Efficacy and Safety of Enzyme Replacement Therapies Avalglucosidase Alfa and Alglucosidase Alfa Administered Every Other Week in Patients With Late-onset Pompe Disease Who Have Not Been Previously Treated for Pompe Disease
Acronym: COMET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC14028; 2016-000942-77 (EudraCT Number); U1111-1178-4806 (Other: WHO universal trial number)
Record Dates: First submitted 2016-05-23; First posted 2016-05-25 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Glycogen Storage Disease Type II;Pompe's Disease
MeSH Terms: interventions — GAA protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- avalglucosidase alfa (GZ402666) (Experimental): Administered intravenously every 2 weeks
  Interventions: Drug: Avalglucosidase alfa (GZ402666)
- alglucosidase alfa (GZ419829) (Active Comparator): Administered intravenously every 2 weeks
  Interventions: Drug: Alglucosidase alfa (GZ419829)

INTERVENTIONS:
Drug: Avalglucosidase alfa (GZ402666) — Pharmaceutical form: powder for concentrate for solution for infusion Route of administration: intravenous
  Arms: avalglucosidase alfa (GZ402666)
Drug: Alglucosidase alfa (GZ419829) — Pharmaceutical form: powder for concentrate for solution for infusion Route of administration: intravenous
  Other Names: Myozyme; Lumizyme
  Arms: alglucosidase alfa (GZ419829)

SUMMARY:
Primary Objective:

To determine the effect of avalglucosidase alfa treatment on respiratory muscle strength measured by percent (%) predicted forced vital capacity (FVC) in the upright position, as compared to alglucosidase alfa.

Secondary Objective:

To determine the safety and effect of avalglucosidase alfa treatment on functional endurance (6-minute walk test, inspiratory muscle strength (maximum inspiratory pressure), expiratory muscle strength (maximum expiratory pressure), lower extremity muscle strength (hand-held dynamometry), motor function (Quick Motor Function Test), and health-related quality of life (Short Form-12).

DETAILED DESCRIPTION:
The duration of the study per participant will be up to approximately 6 years that will consist of a 14-day screening period (may be extended up to 8 weeks in pre-specified situations), a 49-week blinded treatment period (except for the subgroup of pediatric patients aged 3 to less than (<) 18 years enrolling directly in the open-label long-term follow-up phase), a 240-week open-label treatment period, and a 4-week post-treatment observation period.

ELIGIBILITY:
Inclusion criteria :

* The participant has confirmed acid alpha-glucosidase (GAA) enzyme deficiency from any tissue source and/or 2 confirmed GAA gene mutations.
* The participant must provide signed, informed consent prior to performing any study related procedures. Consent of a legally authorized guardian(s) is (are) required for legally minor participant as defined by local regulation. If the participant is legally minor, signed written consent shall be obtained from parent(s)/legal guardian and assent obtained from participants, if applicable.

Exclusion criteria:

* The participant is <3 years of age.
* The participant has known Pompe specific cardiac hypertrophy.
* The participant is wheelchair dependent.
* The participant is not able to ambulate 40 meters (approximately 130 feet) without stopping and without an assistive device.
* The participant requires invasive-ventilation (non-invasive ventilation is allowed).
* The participant is not able to successfully perform repeated forced vital capacity (FVC) measurements in upright position of greater than or equal to 30% predicted and less than or equal to 85% predicted.
* The participant (and participant's legal guardian if participant is legally minor as defined by local regulation) is (are) not able to comply with the clinical protocol.
* The participant has had previous treatment with alglucosidase alfa or any investigational therapy for Pompe disease.
* The participant has prior or current use of immune tolerance induction therapy.
* The participant, if female and of childbearing potential, has a positive pregnancy test (beta-human chorionic gonadotropin) at baseline.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (69):
- United States (21):
  - Investigational Site Number 8400015, Phoenix, Arizona
  - Investigational Site Number 8400020, Los Angeles, California
  - Investigational Site Number 8400011, Orange, California
  - Investigational Site Number 8400017, Stanford, California
  - Investigational Site Number 8400016, Gainesville, Florida
  - Investigational Site Number 8400007, Decatur, Georgia
  - Investigational Site Number 8400023, Chicago, Illinois
  - Investigational Site Number 8400002, Iowa City, Iowa
  - Investigational Site Number 8400012, Kansas City, Kansas
  - Investigational Site Number 8400010, Boston, Massachusetts
  - Investigational Site Number 8400001, Detroit, Michigan
  - Investigational Site Number 8400019, Minneapolis, Minnesota
  - Investigational Site Number 8400026, Great Neck, New York
  - Investigational Site Number 8400008, Valhalla, New York
  - Investigational Site Number 8400006, Durham, North Carolina
  - Investigational Site Number 8400009, Cincinnati, Ohio
  - Investigational Site Number 8400014, Portland, Oregon
  - Investigational Site Number 8400025, Pittsburgh, Pennsylvania
  - Investigational Site Number 8400018, Salt Lake City, Utah
  - Investigational Site Number 8400005, Fairfax, Virginia
  - Investigational Site Number 8400024, Morgantown, West Virginia
- Investigational Site Number 0320001, Caba, Argentina
- Investigational Site Number 0360001, Auchenflower, Australia
- Investigational Site Number 0400001, Vienna, Austria
- Belgium (2):
  - Investigational Site Number 0560003, Brussels
  - Investigational Site Number 0560001, Leuven
- Brazil (2):
  - Investigational Site Number 0760004, Brasília
  - Investigational Site Number 0760001, São Paulo
- Canada (2):
  - Investigational Site Number 1240003, Hamilton
  - Investigational Site Number 1240002, Montreal
- Investigational Site Number 2030001, Prague, Czechia
- Investigational Site Number 2080003, København Ø, Denmark
- France (8):
  - Investigational Site Number 2500008, Angers
  - Investigational Site Number 2500007, Bordeaux
  - Investigational Site Number 2500011, Brest
  - Investigational Site Number 2500004, Bron
  - Investigational Site Number 2500010, Clermont-Ferrand
  - Investigational Site Number 2500005, Lille
  - Investigational Site Number 2500006, Marseille
  - Investigational Site Number 2500001, Paris
- Germany (4):
  - Investigational Site Number 2760006, Bochum
  - Investigational Site Number 2760001, Mainz
  - Investigational Site Number 2760003, München
  - Investigational Site Number 2760002, Münster
- Investigational Site Number 3480001, Budapest, Hungary
- Italy (5):
  - Investigational Site Number 3800006, Brescia
  - Investigational Site Number 3800001, Messina
  - Investigational Site Number 3800002, Milan
  - Investigational Site Number 3800007, Napoli
  - Investigational Site Number 3800003, Torino
- Investigational Site Number 3920002, Kodaira-Shi, Japan
- Investigational Site Number 4840001, México, Mexico
- Investigational Site Number 5280001, Rotterdam, Netherlands
- Investigational Site Number 6160001, Warsaw, Poland
- Investigational Site Number 6200001, Braga, Portugal
- Investigational Site Number 6430001, Moscow, Russia
- South Korea (2):
  - Investigational Site Number 4100001, Seoul
  - Investigational Site Number 4100002, Seoul
- Spain (2):
  - Investigational Site Number 7240002, Barcelona
  - Investigational Site Number 7240003, Barcelona
- Investigational Site Number 7560002, Zurich, Switzerland
- Investigational Site Number 1580001, Taipei, Taiwan
- Turkey (Türkiye) (2):
  - Investigational Site Number 7920001, Ankara
  - Investigational Site Number 7920002, Istanbul
- United Kingdom (5):
  - Investigational Site Number 8260005, Birmingham
  - Investigational Site Number 8260002, Cambridge
  - Investigational Site Number 8260001, London
  - Investigational Site Number 8260004, Newcastle upon Tyne
  - Investigational Site Number 8260003, Salford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kishnani PS, Diaz-Manera J, Illarioshkin S, van der Ploeg AT, Clemens PR, Day JW, Toscano A, Kushlaf H, Ladha S, Attarian S, Carvalho G, Kostera-Pruszczyk A, Erdem-Ozdamar S, Goker-Alpan O, Mozaffar T, Straub V, Roberts M, Haack KA, Huynh-Ba O, Tammireddy S, Periquet M, Thibault N, Zhou T, Dimachkie MM, Schoser B; COMET Investigator Group. Efficacy and safety of avalglucosidase alfa in patients with late-onset Pompe disease after 145 weeks of treatment during the COMET trial. J Neurol. 2025 Aug 16;272(9):581. doi: 10.1007/s00415-025-13266-y. PMID 40817977
- [Derived] Dimachkie MM, Kishnani PS, Ivanescu C, Flore G, Gwaltney C, van der Beek NAME, Hamed A, An Haack K, Pollissard L, Baranowski E, Sparks SE, DasMahapatra P; for COMET Study Group. Measurement Properties of 2 Novel PROs, the Pompe Disease Symptom Scale and Pompe Disease Impact Scale, in the COMET Study. Neurol Clin Pract. 2023 Oct;13(5):e200181. doi: 10.1212/CPJ.0000000000200181. Epub 2023 Aug 8. PMID 37559825
- [Derived] Kishnani PS, Diaz-Manera J, Toscano A, Clemens PR, Ladha S, Berger KI, Kushlaf H, Straub V, Carvalho G, Mozaffar T, Roberts M, Attarian S, Chien YH, Choi YC, Day JW, Erdem-Ozdamar S, Illarioshkin S, Goker-Alpan O, Kostera-Pruszczyk A, van der Ploeg AT, An Haack K, Huynh-Ba O, Tammireddy S, Thibault N, Zhou T, Dimachkie MM, Schoser B; COMET Investigator Group. Efficacy and Safety of Avalglucosidase Alfa in Patients With Late-Onset Pompe Disease After 97 Weeks: A Phase 3 Randomized Clinical Trial. JAMA Neurol. 2023 Jun 1;80(6):558-567. doi: 10.1001/jamaneurol.2023.0552. PMID 37036722
- [Derived] Diaz-Manera J, Kishnani PS, Kushlaf H, Ladha S, Mozaffar T, Straub V, Toscano A, van der Ploeg AT, Berger KI, Clemens PR, Chien YH, Day JW, Illarioshkin S, Roberts M, Attarian S, Borges JL, Bouhour F, Choi YC, Erdem-Ozdamar S, Goker-Alpan O, Kostera-Pruszczyk A, Haack KA, Hug C, Huynh-Ba O, Johnson J, Thibault N, Zhou T, Dimachkie MM, Schoser B; COMET Investigator Group. Safety and efficacy of avalglucosidase alfa versus alglucosidase alfa in patients with late-onset Pompe disease (COMET): a phase 3, randomised, multicentre trial. Lancet Neurol. 2021 Dec;20(12):1012-1026. doi: 10.1016/S1474-4422(21)00241-6. PMID 34800399

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 69 centers in 26 countries. A total of 149 participants were screened between 02 November 2016 and 22 March 2019, of which 100 participants were enrolled and randomized (1:1 ratio) to receive avalglucosidase alfa or alglucosidase alfa. A total of 48 participants were screen failure mainly due to meeting exclusion criteria. 1 pediatric participant entered open-label treatment period directly.
Pre-assignment Details: Randomization was stratified by baseline percent (%) predicted forced vital capacity (FVC): less than (<) 55% or greater than or equal to (>=) 55%, gender, age (<18 years and >=18 years), and country (Japan or ex-Japan). Data reported based on study completion date, i.e. 31 May 2023.
Groups:
- Avalglucosidase Alfa: Avalglucosidase alfa 20 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks (q2w) up to Week 49 in blinded treatment period (also known as primary analysis period [PAP]); followed by same treatment from Week 50 to 289 in an open-label avalglucosidase alfa long-term follow-up phase.
- Alglucosidase Alfa in PAP Then Avalglucosidase Alfa in Open-label: Alglucosidase alfa, 20 mg/kg IV infusion q2w up to Week 49 in blinded treatment period (also known as PAP); followed by avalglucosidase alfa 20 mg/kg IV infusion q2w treatment from Week 50 to 289 in an open-label avalglucosidase alfa long-term follow-up phase.
- Avalglucosidase Alfa in Open-label Only: One participant included directly in the open-label long-term period (Week 50 to 289) and received avalglucosidase alfa 20 mg/kg IV infusion q2w throughout the treatment period.
Period: Blinded Treatment Period: up to Week 49
Arm/Group | Avalglucosidase Alfa | Alglucosidase Alfa in PAP Then Avalglucosidase Alfa in Open-label | Avalglucosidase Alfa in Open-label Only
Started (Randomized and treated participants.) | 51 | 49 | 0
Safety Population (Included participants who received at least 1 infusion in blinded treatment period (also known as PAP) and were analyzed according to the treatment received.) | 51 | 49 | 0
Completed | 51 | 44 | 0
Not Completed | 0 | 5 | 0
Not completed — Adverse Event | 0 | 4 | 0
Not completed — Other | 0 | 1 | 0
Period: Open-label Long-term: Week 50 to 289
Arm/Group | Avalglucosidase Alfa | Alglucosidase Alfa in PAP Then Avalglucosidase Alfa in Open-label | Avalglucosidase Alfa in Open-label Only
Started | 51 | 44 | 1
Safety Population (Included participants who received at least 1 infusion in open-label long-term phase and were analyzed according to the treatment received.) | 51 | 44 | 1
Completed | 44 | 36 | 1
Not Completed | 7 | 8 | 0
Not completed — Adverse Event | 2 | 3 | 0
Not completed — Poor compliance to protocol | 0 | 1 | 0
Not completed — Other | 5 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all randomized participants who had received at least 1 infusion (partial or total) and were analyzed according to the treatment arm allocated by randomization.
Groups:
- Avalglucosidase Alfa: Avalglucosidase alfa, 20 mg/kg IV infusion q2w up to Week 49 in blinded treatment period (also known as PAP); followed by same treatment from Week 50 to 289 in an open-label avalglucosidase alfa long-term follow-up phase.
- Total: Total of all reporting groups
Arm/Group | Avalglucosidase Alfa | Alglucosidase Alfa in PAP Then Avalglucosidase Alfa in Open-label | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (14.5) | 50.3 (13.7) | 48.1 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 27 | 25 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 47 | 47 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Percent Predicted Forced Vital Capacity (FVC) in Upright Position [Mean (Standard Deviation); unit: percent predicted FVC] — FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position.
  percent predicted FVC | 62.5 (14.4) | 61.6 (12.4) | 62.1 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: PAP: Change From Baseline in Percent Predicted FVC in Upright Position at Week 49
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC is the volume of air (in liters) that can be forcibly blown out after full inspiration in the upright position. Least square (LS) mean and standard error (SE) were derived from mixed model for repeated measure (MMRM) model with baseline FVC [percent (%) predicted, as continuous], sex, age (in years at baseline), treatment group, visit, interaction term between treatment group and visit as fixed effects. Percent of predicted FVC = (actual FVC measurement)/(predicted value of FVC) * 100. After non-inferiority (NI) testing, a test for superiority of avalglucosidase alfa versus alglucosidase alfa was performed with an overall 2-sided 5% level of significance.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent predicted FVC
Groups:
- PAP: Avalglucosidase Alfa: Avalglucosidase alfa, 20 mg/kg IV infusion q2w up to Week 49 in blinded treatment period (also known as PAP).
- PAP: Alglucosidase Alfa: Alglucosidase alfa, 20 mg/kg IV infusion q2w up to Week 49 in blinded treatment period (also known as PAP).
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
percent predicted FVC | 2.89 (0.88) | 0.46 (0.93)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; Analysis performed using MMRM model with baseline FVC (% predicted, as continuous), sex, age (in years at baseline), treatment group, visit, interaction term between treatment group and visit as fixed effects; Test type: Non-Inferiority — NI was demonstrated if the lower bound of the 2-sided 95% confidence interval (CI) for the difference of avalglucosidase alfa minus alglucosidase alfa was greater than (>) -1.1; p = 0.0074, mixed model for repeated measures; LS mean difference = 2.43, 95% CI 2-sided [-0.13 to 4.99], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — A test for superiority of avalglucosidase alfa versus alglucosidase alfa was performed with an overall 5% level of significance; p = 0.0626, mixed model for repeated measures — Threshold for significance at <0.05 level

2. Secondary Outcome: PAP: Change From Baseline in Total Distance Walked During Six-minute Walk Test (6MWT) at Week 49
Description: 6MWT was a standardized test that measured the distance (in meters) covered by the participant by walking on a flat, hard surface in a period of a 6-minute walk. Mean distance walked gives an indication of functional endurance. The greater the distance (that a participant could walk in 6 minutes), the greater the endurance. LS mean and SE were derived from MMRM model with baseline FVC (% predicted) and baseline 6MWT (distance walked in meter), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
meters | 32.21 (9.93) | 2.19 (10.40)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; LS mean difference was derived from MMRM model with baseline FVC (% predicted) and baseline 6MWT (distance walked in meter), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Superiority — Per the protocol-defined statistical test strategy for multiplicity adjustment, and since superiority was narrowly missed for FVC % predicted, superiority testing for the secondary outcome measure couldn't be performed; p = 0.0405, mixed model for repeated measures; LS mean difference = 30.01, 95% CI 2-sided [1.33 to 58.69], Standard Error of Mean 14.43

3. Secondary Outcome: PAP: Change From Baseline in Percent Predicted Maximal Inspiratory Pressure (MIP) in Upright Position at Week 49
Description: MIP is a quick and non-invasive test to measure strength of inspiratory muscles, primarily diaphragm, and allows for assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MIP refers to how much air pressure force an individual creates by inhaling through the mouth as hard as possible. LS mean and SE were derived from MMRM model for MIP % predicted adjusted for MIP % predicted at baseline, age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent predicted MIP
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
percent predicted MIP | 0.17 (3.60) | -2.96 (3.79)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; LS mean difference was derived from MMRM model for MIP % predicted adjusted for MIP % predicted at baseline, age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.5522, mixed model for repeated measures; LS mean difference = 3.13, 95% CI 2-sided [-7.31 to 13.57], Standard Error of Mean 5.24

4. Secondary Outcome: PAP: Change From Baseline in Percent Predicted Maximal Expiratory Pressure (MEP) in Upright Position at Week 49
Description: MEP is a quick and non-invasive test to measure strength of expiratory muscles, primarily diaphragm, and allows for assessment of ventilatory failure, restrictive lung disease and respiratory muscle strength. MEP is the greater pressure generated during maximal expiration. LS mean and SE were derived from MMRM model for MEP % predicted adjusted for MEP % predicted at baseline, age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: percent predicted MEP
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
percent predicted MEP | 3.02 (3.87) | 4.95 (4.07)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; LS mean difference was derived from MMRM model for MEP % predicted adjusted for MEP % predicted at baseline, age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.7321, mixed model for repeated measures; LS mean difference = -1.94, 95% CI 2-sided [-13.17 to 9.29], Standard Error of Mean 5.64

5. Secondary Outcome: PAP: Change From Baseline in Lower Extremity Muscle Strength at Week 49 as Assessed by Hand-Held Dynamometry (HHD)
Description: HHD: a portable method for strength quantitation. To complete a make test, participant exerted maximal force against dynamometer with gradual increase in force and completed isometric hold for 4-5 seconds. Muscle strengths were collected in Newton. Every muscle group (hip: flexion, extension, abduction; knee: flexion, extension and ankle dorsiflexion) were measured 2 times and highest value was reported. Summary score was sum of 12 measurements (2 measurements per muscle group) from 6 muscle groups on each side (left and right). An increase from Baseline was reflective of increased muscle strength, whereas a decrease from Baseline was reflective of decreased muscle strength. LS mean and SE were derived from MMRM model for HHD lower extremity muscle strength composite score adjusted for summary HHD lower extremity score at baseline, baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: Newton
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
Newton | 260.69 (46.07) | 153.72 (48.54)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; LS mean difference was derived from MMRM model for HHD lower extremity muscle strength composite score adjusted for summary HHD lower extremity score at baseline, baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.1150, mixed model for repeated measures; LS mean difference = 106.97, 95% CI 2-sided [-26.56 to 240.50], Standard Error of Mean 67.17

6. Secondary Outcome: PAP: Change From Baseline in Quick Motor Function Test (QMFT) Total Scores at Week 49
Description: The QMFT was an observer administered test to evaluate changes in motor function. QMFT comprised of 16 items specifically difficult for participants with Pompe disease. Each item was scored separately on a 5-point ordinal scale (ranged from 0 to 4, higher score indicated better outcome). Total QMFT score was obtained by adding the scores of all items and ranged from 0 (unable to perform motor function tests) to 64 (normal muscle function), higher score represented better outcome. LS mean and SE were derived from MMRM models adjusted for total QMFT score at baseline, baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
scores on a scale | 3.98 (0.63) | 1.89 (0.69)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; LS mean difference was derived from MMRM models adjust for total QMFT score at baseline, baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Other — No formal testing of additional secondary endpoint of QMFT; p = 0.0288, mixed model for repeated measures — Nominal p-value; LS mean difference = 2.08, 95% CI 2-sided [0.22 to 3.95], Standard Error of Mean 0.94

7. Secondary Outcome: PAP: Change From Baseline in 12-Item Short-Form Health Survey (SF-12): Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores at Week 49
Description: SF-12, a 12 item-questionnaire, used to assess health-related quality of life in participants aged >=18 years at screening/baseline. SF-12 consisted of 12 items, which were categorized into eight domains (subscales) of functioning and well-being: physical functioning, role-physical, role emotional, mental health, bodily pain, general health, vitality and social functioning, with each domain score ranged from 0 (poor health) to 100 (better health), higher scores indicated good health condition. These eight domains were further summarized into 2 summary scores, PCS and MCS. The score range for each of these 2 summary scores was from 0 (poor health) to 100 (better health), higher scores indicated a better health-related quality of life. LS mean and SE were derived from MMRM models adjusted for baseline score (PCS or MCS), baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 49
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 50 | 49
scores on a scale
  PCS score | 2.37 (0.99) | 1.60 (1.07)
  MCS score | 2.88 (1.22) | 0.76 (1.32)
Statistical Analysis 1: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; The MMRM models adjust for baseline score (PCS), baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Other — No formal testing of additional secondary endpoint of SF-12; p = 0.5996, mixed model for repeated measures; Score difference = 0.77, 95% CI 2-sided [-2.13 to 3.67], Standard Error of Mean 1.46
Statistical Analysis 2: Comparison: PAP: Avalglucosidase Alfa vs PAP: Alglucosidase Alfa; The MMRM models adjust for baseline score (MCS), baseline FVC (% predicted), age (in years, at baseline), gender, treatment group, visit, and treatment-by-visit interaction as fixed effects; Test type: Other — No formal testing of additional secondary endpoint of SF-12; p = 0.2427, mixed model for repeated measures; Score difference = 2.12, 95% CI 2-sided [-1.46 to 5.69], Standard Error of Mean 1.80

8. Secondary Outcome: PAP: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Infusion-Associated Reactions (IARs)
Description: AE: any untoward medical occurrence in participant who took study drug and not necessarily have to had causal relationship with treatment. TEAEs: AEs that developed/worsened in grade/became serious during TEAE period in PAP (from time of 1st treatment date to last treatment date+4 weeks for participants who didn't receive any treatment in open-label or to time just prior to 1st treatment in open-label for participants who received treatment in open-label). Protocol-defined IARs: AE of special interest (AESIs) that occurred during either infusion/observation period following infusion which were deemed to be related/possibly related to study drug. Algorithm-defined IARs: any TEAE meeting either 1 of 2 criteria: 1) event occurred from start to end of infusion + 24 hours, considered related to study drug, 2) If AE time component missed, compare AE start date with infusion start and end date. If AE start date was between infusion start and end date + 1 day and it was related to study drug.
Time Frame: From Baseline up to Week 49
Population: Analysis was performed on safety population which included participants who had received at least 1 infusion (partial or total) and were analyzed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 49
Participants
  Any TEAE | 44 | 45
  Any Protocol-defined IARs | 13 | 16
  Any Algorithm-defined IARs | 15 | 20

9. Secondary Outcome: Open-label Period: Number of Participants With TEAEs and IARs
Description: AE: any untoward medical occurrence in a participant who received study drug and did not necessarily have to had a causal relationship with treatment. TEAEs in open-label: AEs that developed/worsened in grade/became serious during TEAE period in open-label (from time of 1st open-label treatment to last treatment date + 4 weeks). Protocol-defined IARs: defined as AESIs that occurred during either infusion/observation period following infusion which were deemed to be related/possibly related to study drug. Algorithm-defined IARs: any TEAE meeting either 1 of 2 criteria: 1) event occurred from start to end of infusion plus 24 hours, considered related to study drug, 2) If AE time component missed, compare AE start date with infusion start and end date. If AE start date was between infusion start and end date plus 1 day and it was related to study drug.
Time Frame: Week 50 to 289 in open-label long-term period
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Avalglucosidase Alfa-Open-label After Avalglucosidase Alfa-PAP; Avalglucosidase Alfa-Open-label After Alglucosidase Alfa-PAP: Avalglucosidase alfa 20 mg/kg IV infusion q2w from Week 50 up to 289 based on product approval status in an open-label avalglucosidase alfa long-term follow-up phase.
Arm/Group | Avalglucosidase Alfa-Open-label After Avalglucosidase Alfa-PAP | Avalglucosidase Alfa-Open-label After Alglucosidase Alfa-PAP | Avalglucosidase Alfa in Open-label Only
Number analyzed (Participants) | 51 | 44 | 1
Participants
  Any TEAE | 51 | 43 | 1
  Any Protocol-defined IARs | 12 | 22 | 0
  Any Algorithm-defined IARs | 16 | 24 | 0

10. Secondary Outcome: PAP: Percentage of Participants With Treatment-Emergent Antidrug Antibodies (ADA) Response
Description: ADA response categories: 1) Treatment-induced: ADAs developed following administration of the study drug. If the baseline ADA sample was missing or non-reportable and at least one reportable on-treatment ADA sample was available, the baseline sample was considered as "negative". 2) Treatment-boosted: Pre-existing ADAs that were boosted at least two titer steps from baseline (i.e., 4 fold increase in titers) following administration of the study drug (any time after the first drug administration). 3) Treatment emergent: combination of treatment induced and treatment boosted.
Time Frame: From Baseline up to Week 49
Population: Analysis was performed on ADA evaluable population which consisted of participants who had received at least 1 infusion (partial or total) and had at least one ADA sample taken post-baseline after drug administration that was appropriate for ADA testing with a reportable result.
Measure: Number; unit: percentage of participants
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa
Number analyzed (Participants) | 51 | 48
percentage of participants
  Treatment-Induced | 95.9 | 95.7
  Treatment-boosted ADA | 100 | 100
  Treatment emergent ADA | 96.1 | 95.8

ADVERSE EVENTS:
Time Frame: Up to Week 49 in PAP and from Week 50 to 289 in open-label long-term period
Description: AEs and deaths: TEAEs that developed/worsened in grade/became serious during 'TEAE period' (PAP: from first treatment date to last treatment date+4 weeks for participants not exposed to treatment in open-label or to time just prior to first dose in open-label for those exposed to open-label [time from first study drug to last dose+4 weeks]). Safety population.
Groups:
- PAP: Avalglucosidase Alfa: Avalglucosidase alfa 20 mg/kg IV infusion q2w up to Week 49 in blinded treatment period (also known as PAP).
- PAP: Alglucosidase Alfa: Alglucosidase alfa 20 mg/kg IV infusion q2w up to Week 49 in blinded treatment period (also known as PAP).
- Open-label: Avalglucosidase Alfa: Included all subjects who received avalglucosidase alfa, 20 mg/kg IV infusion q2w from Week 50 up to 289 based on product approval status in an open-label avalglucosidase alfa long-term follow-up phase.
- Open-label: Alglucosidase Alfa-PAP Then Avalglucosidase Alfa: Included all subjects who received avalglucosidase alfa 20 mg/kg IV infusion q2w treatment from Week 50 up to 289 based on product approval status in an open-label avalglucosidase alfa long-term follow-up phase.
Arm/Group | PAP: Avalglucosidase Alfa | PAP: Alglucosidase Alfa | Open-label: Avalglucosidase Alfa | Open-label: Alglucosidase Alfa-PAP Then Avalglucosidase Alfa
All-Cause Mortality (participants affected / at risk) | 0/51 | 1/49 | 0/52 | 2/44
Serious Adverse Events (participants affected / at risk) | 8/51 | 12/49 | 14/52 | 14/44
Other Adverse Events (participants affected / at risk) | 40/51 | 44/49 | 50/52 | 40/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: Avalglucosidase Alfa (N=51) | PAP: Alglucosidase Alfa (N=49) | Open-label: Avalglucosidase Alfa (N=52) | Open-label: Alglucosidase Alfa-PAP Then Avalglucosidase Alfa (N=44)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6)
Brain Stem Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar Ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed Level Of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Moyamoya Disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diaphragmatic Paralysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (4) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Tongue Oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glycogen Storage Disease Type Ii (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viiith Nerve Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PAP: Avalglucosidase Alfa (N=51) | PAP: Alglucosidase Alfa (N=49) | Open-label: Avalglucosidase Alfa (N=52) | Open-label: Alglucosidase Alfa-PAP Then Avalglucosidase Alfa (N=44)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 4 (4)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 16 (17) | 9 (9)
Cystitis (Infections and infestations) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 10 (11) | 3 (4) | 4 (4) | 4 (5)
Nasopharyngitis (Infections and infestations) | 12 (15) | 12 (17) | 15 (23) | 13 (27)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (5) | 2 (2) | 3 (4) | 8 (10)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 1 (4) | 8 (10) | 3 (9)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 5 (5) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6) | 3 (14) | 6 (8) | 3 (4)
Headache (Nervous system disorders) | 11 (32) | 16 (102) | 12 (42) | 17 (220)
Paraesthesia (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 3 (12) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Ocular Hyperaemia (Eye disorders) | 1 (3) | 1 (1) | 3 (4) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Flushing (Vascular disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (3)
Hypertension (Vascular disorders) | 1 (2) | 3 (5) | 7 (21) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 4 (7) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (3) | 3 (5)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 2 (2) | 2 (2)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (8) | 2 (6) | 4 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (8) | 4 (6)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (4) | 2 (2) | 3 (6) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (9) | 8 (9) | 7 (15) | 14 (19)
Dyspepsia (Gastrointestinal disorders) | 3 (9) | 3 (5) | 2 (2) | 3 (9)
Nausea (Gastrointestinal disorders) | 6 (8) | 7 (15) | 12 (16) | 7 (22)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (3) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (3) | 3 (4) | 6 (7)
Erythema (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (7) | 3 (4) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (11) | 3 (3) | 11 (51)
Rash (Skin and subcutaneous tissue disorders) | 2 (11) | 4 (4) | 4 (8) | 8 (16)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (5) | 5 (12) | 4 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 8 (11) | 13 (27) | 13 (29)
Back Pain (Musculoskeletal and connective tissue disorders) | 12 (15) | 5 (7) | 11 (13) | 10 (20)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 4 (7) | 5 (8)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (6) | 1 (1) | 3 (5)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (117)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (15) | 7 (12) | 6 (12) | 10 (22)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (5) | 3 (4) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 8 (9) | 8 (15) | 10 (29) | 9 (19)
Dysuria (Renal and urinary disorders) | 2 (4) | 0 (0) | 0 (0) | 3 (3)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Chills (General disorders) | 1 (1) | 2 (6) | 4 (13) | 5 (13)
Fatigue (General disorders) | 9 (11) | 7 (27) | 4 (8) | 9 (75)
Influenza Like Illness (General disorders) | 2 (4) | 0 (0) | 3 (8) | 1 (1)
Infusion Site Extravasation (General disorders) | 0 (0) | 3 (3) | 2 (2) | 5 (8)
Oedema Peripheral (General disorders) | 3 (4) | 3 (3) | 5 (7) | 4 (4)
Pain (General disorders) | 2 (3) | 5 (13) | 3 (5) | 6 (14)
Peripheral Swelling (General disorders) | 1 (3) | 3 (3) | 1 (1) | 5 (6)
Pyrexia (General disorders) | 2 (2) | 4 (4) | 8 (10) | 6 (11)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 3 (3) | 1 (1) | 2 (2)
Blood Pressure Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 5 (7) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 7 (12) | 10 (13) | 10 (28) | 8 (21)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/41/NCT02782741/Prot_002.pdf
  • Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT02782741/SAP_003.pdf